CLINICAL TRIAL: NCT03909282
Title: A Randomized Phase II Study Comparing Surgical Excision Versus Neoadjuvant Radiotherapy Followed by Delayed Surgical Excision of Ductal Carcinoma In Situ (NORDIS)
Brief Title: Surgical Excision vs Neoadjuvant Radiotherapy+Delayed Surgical Excision of Ductal Carcinoma
Acronym: NORDIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-46373; BRS0096 (Other: OnCore); NCI-2019-02516 (Other: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2019-04-02; First posted 2019-04-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Ductal Breast Carcinoma in Situ
Keywords: Ductal Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast | interventions — Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Surgical Excision (Active Comparator): Surgical excision of ductal carcinoma
  Interventions: Procedure: Lumpectomy
- Neoadjuvant partial breast irradiation (Experimental): Partial breast irradiation will be delivered once a day for 5 days before surgery. The planned daily dose is 6 Gy.
  Interventions: Procedure: Lumpectomy; Radiation: Partial breast irradiation prior to surgery

INTERVENTIONS:
Procedure: Lumpectomy — Standard of Care surgery for DCIS (either lumpectomy or mastectomy)
  Other Names: Mastectomy
Radiation: Partial breast irradiation prior to surgery — Partial breast irradiation (PBI) will be delivered once aday for 5 days. The planned daily dose is 6 Gy prior to surgery (neo adjuvant)
  Arms: Neoadjuvant partial breast irradiation

SUMMARY:
The purpose of this pilot study is to compare by pathological findings surgical excision versus neoadjuvant radiotherapy followed by delayed surgical excision of ductal carcinoma in situ (DCIS)

DETAILED DESCRIPTION:
There will be measurable histopathological treatment effects identified in Arm 2 cases receiving pre-operative radiation. Results found are expected to assist in designing a more definitive study. Compare pathological findings in individuals with ductal carcinoma in situ (DCIS) who have surgical excision versus neoadjuvant radiotherapy followed by delayed surgical excision.

It is noted that "phase 2" is formally associated with drug studies. Nonetheless, it is however part of the time of this study.

ELIGIBILITY:
Inclusion Criteria

* Core needle biopsy demonstrating DCIS (ductal carcinoma in situ) of non-palpable, image-detected breast abnormality
* Signed and dated IRB-approved written informed consent
* Women 18 years of age or older
* Mammographic calcifications or MRI non-mass enhancement measuring 4 cm or less in greatest dimension, including multifocal disease
* Estrogen receptor positive or negative, progesterone receptor positive or negative DCIS; HER2 positive, negative or unknown DCIS is allowed.
* Diagnostic needle biopsy within 16 weeks of randomization
* Patients must have a biopsy marker placed within the tumor bed confirmed on post biopsy imaging and evidence of residual radiographic abnormality. Confirmation of residual imaging abnormality is required within 6 weeks of randomization.
* Placement of Savi scout optical reflectance marker in tumor bed area as a wireless guide for surgery and for neoRT treatment planning is preferred but not required if anatomic metallic markers are sufficient for radiation planning. Placement does not have to occur before randomization. Additionally, wire localization before surgery is permissible.
* Planned lumpectomy. Mastectomy will be acceptable if lumpectomy fails by virtue of involved margins or size of lesion, or patient chooses this approach after randomization
* Radiation Oncologist to ascertain feasibility of PBI prior to randomization - based on their estimation that 30% or less of the breast volume will be encompassed in the radiation fields
* Patients who had a prior contralateral invasive or non-invasive (DCIS) cancer are eligible
* ECOG performance status 0, 1, or 2
* Concurrent foci of atypia or lobular carcinoma in situ in the ipsilateral or contralateral breast are allowed

Exclusion Criteria

* Invasive carcinoma on core needle biopsy, including microinvasive carcinoma
* Radiographic extent of DCIS >4.0 cm
* Mass lesion on breast imaging or palpable tumor
* No residual radiographic lesion after diagnostic percutaneous core needle biopsy
* Prior history of ipsilateral invasive or noninvasive breast cancer
* Pregnant or breastfeeding
* Prior ipsilateral breast or chest irradiation
* Multicentric or multifocal DCIS, if extent is > 4cm
* Synchronous contralateral invasive or noninvasive breast cancer
* Pagets' disease of the breast
* Active collagen vascular disease
* Positive axillary lymph nodes
* Not meeting the described criteria for partial breast irradiation during initial clinical evaluation.
* Psychiatric or addictive disorders or other condition, that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or interfere with the interpretation of study results
* Endocrine therapy is not allowed from the time of study randomization to the completion of surgery unless the endocrine therapy is being continued for a contralateral cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-03-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of ductal carcinoma in situ (DCIS) pathologic complete response | 12 weeks
  A DCIS pathologic complete response will be defined as the absence of in situ carcinoma in the surgical resection specimen. The rate of DCIS pathologic complete response (pCR) will be calculated for Arm 1 and Arm 2.

SECONDARY OUTCOMES:
Correlation of ductal carcinoma in situ (DCIS) subtypes with rate of DCIS pathologic complete response to neoadjuvant partial breast irradiation (PBI) | 12 weeks
  Molecular subtypes based on gene expression profiling with therapy response will be corelated.
  • DCIS subtypes will be defined based on grade, estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER2) status as follows:
  * Low/intermediate grade versus high grade
  * ER/PR-negative versus ER/PR-positive
  * HER2-positive versus HER2-negative
Tumor grade comparison of radiation-induced treatment effect pathologically pre- versus post-therapy | 12 weeks
  Tumor grade (grade 1, 2, 3) will be compared pre- and post-therapy.
Nuclear atypia comparison of radiation-induced treatment effect pathologically pre- versus post-therapy | 12 weeks
  Degree of nuclear atypia (low, intermediate, high) will be compared pre- and post-therapy.
Percent tumor necrosis comparison of radiation-induced treatment effect pathologically pre- versus post-therapy | 12 weeks
  Percent tumor necrosis (0-100%) will be quantified on the basis of percentage of overall residual tumor area and compared pre- and post-treatment.
Tumor cellularity comparison of radiation-induced treatment effect pathologically pre- versus post-therapy | 12 weeks
  Tumor cellularity (0-100%) will be quantified on the basis of percentage of overall residual tumor area and compared pre- and post-treatment.
Proportion of subjects experiencing a wound complication on Arm 1 compared to Arm 2 | 12 weeks
  Wound complications and healing will be monitored in both arms.The following events will be considered wound complications: wound dehiscence, hematoma requiring intervention, seroma requiring drainage, skin necrosis requiring resection, cellulitis requiring antibiotic therapy.
Correlation of post-radiation imaging characteristics with pathologic findings | 12 weeks
  Mammography obtained prior to surgical resection in Arm 2 patients will be assessed for the presence or absence of a residual mammographic abnormality, the size in mm of the residual mammographic abnormality and the longest span in mm of residual calcification and will be compared to the pathologic presence or absence of residual tumor, size in mm of the pathologic residual DCIS and whether the residual calcification is associated with pathologic residual DCIS.
Rate of invasive carcinoma comparison in Arm 1 to Arm 2 | 12 weeks
  Rate of pathologic residual invasive carcinoma will be assessed in Arm 1 and Arm 2.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Wapnir, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No